CLINICAL TRIAL: NCT04766411
Title: Recovery Kinetics After Different Sprint Training Protocols
Brief Title: Recovery Kinetics After Different Sprint Training Protocols (STRecovery)
Acronym: STRecovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Chariklia K. Deli, Assistant Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: Sprint training-Recovery Study
Record Dates: First submitted 2021-02-11; First posted 2021-02-23 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Sprint Training
Keywords: sprint training; muscle damage; muscle performance; neuromuscular fatigue; recovery
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Unresisted sprint training (Experimental): Participants will perform an acute training bout of unresisted sprints.
  Interventions: Other: Unresisted sprint training
- Resisted sprint training with load equal to 10% of body weight (Experimental): Participants will perform an acute training bout of resisted sprints with load equal to 10% of body weight.
  Interventions: Other: Resisted sprint training with load equal to 10% of body weight
- Resisted sprint training with load equal to 20% of body weight (Experimental): Participants will perform an acute training bout of resisted sprints with load equal to 20% of body weight.
  Interventions: Other: Resisted sprint training with load equal to 20% of body weight
- Control trial (Experimental): Participants will perform no training protocol. They will only perform all the measurements.
  Interventions: Other: Control trial

INTERVENTIONS:
Other: Unresisted sprint training — Particiapants will perform:
  2 sets of 3 x 20m sprint
  1 set of 3 x 30m sprint
  Arms: Unresisted sprint training
Other: Resisted sprint training with load equal to 10% of body weight — Particiapants will perform:
  2 sets of 3 x 20m sprint
  1 set of 3 x 30m sprint
  Arms: Resisted sprint training with load equal to 10% of body weight
Other: Resisted sprint training with load equal to 20% of body weight — Particiapants will perform:
  2 sets of 3 x 20m sprint
  1 set of 3 x 30m sprint
  Arms: Resisted sprint training with load equal to 20% of body weight
Other: Control trial — Participants will not perform any sprint training protocol
  Arms: Control trial

SUMMARY:
Speed is one of the most important physical capacities for many sports, especially those that include speed and power as a major element, and plays a major role on performance. Running speed improvement is one of the most basic components of a sprint and power athlete's training program. One of the most commonly used strategies to improve the initial acceleration phase, is resisted sprint training. Sprinting is performed through the stretch-shortening cycle and highly includes the component of eccentric muscle contraction, which can lead to exercise induced muscle damage (EIMD). This phenomenon includes symptoms such as plasma CK elevation, delayed onset of muscle soreness, reduction in force production and a reduction in agility and speed. However, despite the fact that sprint training can cause EIMD symptoms and a performance reduction the following days, research evidence on the recovery kinetics after sprint training are scarce. However, such information is critical for coaches and athletes, in order to effectively design a training program and incorporate the training components in the training microcycle, to avoid injuries and maximize performance. The aim of the present study is to examine the recovery kinetics of EIMD indices, muscle performance and neuromuscular fatigue, after different sprint training protocols.

DETAILED DESCRIPTION:
Speed is one of the most important physical capacities for many sports, especially those that include speed and power as a major element, and plays a major role on performance. Thus, running speed improvement consists one of the most basic aims of a sprinter's and a power athlete's training program. One of the most commonly used strategies to improve the initial acceleration phase, is resisted sprint training. Evidence suggests that resisted sprint training is more effective in improving acceleration compared to sprint training without additional load. Sprinting is performed through the stretch-shortening cycle, where the pre-activated muscle is first stretched (eccentric action) and then followed by the shortening (concentric) action. Thus, sprint training highly includes the component of eccentric contraction. However, eccentric muscle action, especially when unaccustomed, can lead to exercise-induced muscle damage (EIMD). Although concentric and isometric exercise may also lead to muscle injury, the amount of damage after eccentric muscle contractions is greater. EIMD, amongst others, is accompanied by increased levels of creatine kinase (CK) into the circulation, increased delayed onset of muscle soreness (DOMS), reduction of force production, reduction of agility and speed. Nevertheless, despite the fact that sprint training comprises eccentric muscle actions and consequently can lead to muscle injury and muscle performance reduction during the following days, the recovery kinetics after acute sprint training have not been adequately studied. However, such information is critical for both coaches and athletes to effectively design the training microcycles and incorporate the training components, as well as to reduce injury risk.

The aim of the present study is to examine the recovery kinetics of EIMD indices, muscle performance and neuromuscular fatigue, after different sprint training protocols.

According to a preliminary power analysis (a probability error of 0.05, and a statistical power of 80%), a sample size of 8 - 10 subjects per group was considered appropriate in order to detect statistically meaningful changes between groups.

The study will be performed in a randomized, cross over, repeated measures design. During the first 1st and 2nd visit, all participants will sign an informed consent form after they will be informed about all the benefits and risks of the study and they will fill in and sign a medical history questionnaire. Fasting blood samples will be collected in order to estimate muscle damage concentration markers. Participants will be instructed by a dietitian how to record a 7-days diet recalls to ensure that they do not consume to greater extent nutrients that may affect EIMD and fatigue (e.g. antioxidants, amino acids, etc.) and to ensure that the energy intake during the trials will be the same. Assessment of body mass and body height, body composition, and aerobic capacity (VO2max), will be performed. Running speed of 10 m, 20 m and 30 m sprint will be measured on a track and field stadium. Squat jump and countermovement jump will be performed on a force platform to assess jump height, ground reaction force, peak and mean power, vertical stiffness and peak rate of force development; at the same time, peak and mean normalized EMG during the concentric phase of the squat jump, and during eccentric and concentric phases of the counter movement jump, for the vastus lateralis, biceps femoris, gastrocnemius, and gluteus maximum muscles will be assessed. The peak concentric, eccentric and isometric isokinetic torque of the knee flexors and extensors, in both limbs will be evaluated on an isokinetic dynamometer at 60°/sec. Maximal voluntary isometric contraction (MVIC) of the knee extensors at 65o in both limbs, as well as the fatigue rate during MVIC through the percent drop of peak torque between the first and the last three seconds of a 10-sec MVIC.

During the 3rd visit, participants will be randomly assigned into, and perform one of the four different conditions of the study design: a) unresisted sprint training, b) resisted sprint training with a load of 10% of body weight (BW), c) resisted sprint training with a load of 20% of BW d) control condition. Prior to each experimental protocol, assessment of DOMS in the knee flexors (KF) and extensors (KE) of both limbs, as well as blood lactate assessment will be performed. Additionally, DOMS of KF and KE, running speed at 10 m, 20 m and 30 m sprint, peak concentric, eccentric and isometric isokinetic torque, squat and countermovement jump height, as well as ground reaction force, peak and mean power, vertical stiffness and peak rate of force development during squat and countermovement jump, alongside with peak and mean normalized electromyography (EMG) during the concentric phase of the squat jump, and during eccentric and concentric phases of the counter movement jump, for the vastus lateralis, biceps femoris, gastrocnemius, and tibialis anterior muscles will be assessed immediately after, 24h, 48h and 72h after the end of the trial. MVIC of the knee extensors of both limbs, as well as the fatigue rate during MVIC will also be assessed at 1h, 2h and 3h, as well as 24h, 48h, and 72h after the end of the trial. Blood lactate will also be assessed at 4 min, while creatine kinase at 24h, 48h, and 72h after the end of the trial. The exact above procedures will be repeated by the participants during the remaining three experimental trials (7th - 10th, 11th - 13th, and 14th - 16th visits).

ELIGIBILITY:
Inclusion Criteria:

* Srinters or athletes that comprise sprint training in their training programs
* Absense of musculoskeletal injuries (≥ 6 months)
* Abstence from use of ergogenic supplements or other drugs (≥ 1 month)
* Abstence from participation at exercise with eccentric component (≥ 3 days)
* Abstence from alcohol and energy drings consumption before each experimental trial

Exclusion Criteria:

* Musculoskeletal injuries (≤ 6 months)
* Use of ergogenic supplements or other drugs (≤ 1 month)
* Participation at exercise with eccentric component (≤ 3 days)
* Alcohol and energy drings consumption before the experimental trials

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Changes in Creatine kinase | Baseline (pre), post-, 24 hours post-, 48 hours post-, 72 hours post-trial
  CK will be measured in plasma using a Clinical Chemistry Analyzer with commercially available kits.
Changes in DOMS | Baseline (pre), post-, 24 hours post-, 48 hours post-, 72 hours post-trial
  DOMS of knee extensors and knee flexors of both lower extremities will be measured during palpation of the muscle belly and the distal regionafter performing three repetitions of a full squat.
Changes in blood lactate | Baseline (pre), 4 minutes post-trial
  Lactate will be measured in capillary blood with a hand-portable analyzer.
Changes in 10m sprint time | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  20m sprint time will be measured using light cells Chronojump system.
Changes in 20m sprint time | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  20m sprint time will be measured using light cells Chronojump system.
Changes in 30m sprint time | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  30m sprint time will be measured using light cells Chronojump system.
Changes in squat jump height | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Squat jump height will be measured on a dynamometer using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the data for each leg.
Changes in ground reaction force (GRF) during squat jump | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  GRF during squat jump will be measured on a dynamometer using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the data for each leg.
Changes in peak power during squat jump | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Peak power during squat jump will be measured on a dynamometer using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the data for each leg.
Changes in mean power during squat jump | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Mean power during squat jump will be measured on a dynamometer using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the data for each leg.
Changes in vertical stiffness during squat jump | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Vertical stiffness during squat jump will be measured on a dynamometer using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the data for each leg.
Changes in peak rate of force development (RFD) during squat jump | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  RFD during squat jump will be measured on a dynamometer using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the data for each leg.
Changes in peak normalized EMG during squat jump test | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Electromyography data will be collected wirelessly at 2000Hz using a Myon MA-320 EMG system (Myon AG, Schwarzenberg, Switzerland) for the vastus lateralis, biceps femoris, gastrocnemius, and tibialis anterior muscles during the concentric phase of the squat jump.
Changes in mean normalized EMG during squat jump test. | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Electromyography data will be collected wirelessly at 2000Hz using a Myon MA-320 EMG system (Myon AG, Schwarzenberg, Switzerland) for the vastus lateralis, biceps femoris, gastrocnemius, and tibialis anterior muscles during the concentric phase of the squat jump.
Changes in countermovement jump height | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Countermovement jump height will be measured on a dynamometer using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the data for each leg.
Changes in ground reaction force (GRF) during countermovement jump | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  GRF will be measured on a dynamometer using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the data for each leg.
Changes in peak power during countermovement jump | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Peak power will be measured on a dynamometer using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the data for each leg.
Changes in mean power during countermovement jump | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Mean power will be measured on a dynamometer using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the data for each leg.
Changes in vertical stiffness during countermovement jump | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Vertical stiffnesswill be measured on a dynamometer using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the data for each leg.
Changes in peak rate of force development (RFD) during countermovement jump | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  RFD will be measured on a dynamometer using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the data for each leg.
Changes in peak normalized EMG during countermovement jump test | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Electromyography data will be collected wirelessly at 2000Hz using a Myon MA-320 EMG system (Myon AG, Schwarzenberg, Switzerland) for the vastus lateralis, biceps femoris, gastrocnemius and gluteus maximum muscles during the eccentric and concentric phases of the countermovement jump test.
Changes in mean normalized EMG during countermovement jump test | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Electromyography data will be collected wirelessly at 2000Hz using a Myon MA-320 EMG system (Myon AG, Schwarzenberg, Switzerland) for the vastus lateralis, biceps femoris, gastrocnemius and gluteus maximum muscles during the eccentric and concentric phases of the countermovement jump test.
Changes in peak concentric torque | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Concentric torque of knee extensors and knee flexors will be measured on an isokinetic dynamometer
Changes in peak eccentric torque | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Concentric torque of knee extensors and knee flexors will be measured on an isokinetic dynamometer
Changes in peak isometric torque | Baseline (pre), 24 hours post-, 48 hours post-, 72 hours post-trial
  Concentric torque of knee extensors and knee flexors will be measured on an isokinetic dynamometer
Changes in maximal voluntary isometric contraction (MVIC) | Baseline (pre), 1 hour post-, 2 hours post-, 3 hours post-, 24 hours post-, 48 hours post-, 72 hours post-trial
  MVIC of knee extensors will be measured on an isokinetic dynamometer
Changes in fatigue rate of maximal voluntary isometric contraction (MVIC) | Baseline (pre), 1 hour post-, 2 hours post-, 3 hours post-, 24 hours post-, 48 hours post-, 72 hours post-trial
  Fatigue rate during MVIC will be estimated through the percent drop of peak torque between the first and the last three seconds of a 10-second maximal isometric contaction
Change in field activity during the sprint training protocols | Throughout the sprint training protocols
  Field activity will be continuously recorded during the sprint training protocols using global positioning system (GPS) technology
Change in heart rate during the sprint training protocols | Throughout the sprint training protocols
  Heart rate will be continuously recorded during during the sprint training protocols using heart rate monitors

SECONDARY OUTCOMES:
Body weight | Baseline
  Body weight will be measured on a beam balance with stadiometer
Body height | Baseline
  Body height will be measured on a beam balance with stadiometer
Body mass index (BMI) | Baseline
  BMI will be calculated from the ratio of body mass/ body height squared
Maximal oxygen consumption (VO2max) | Baseline
  Maximal oxygen consumption will be measured by open circuit spirometry via breath by breath method
Body fat | Baseline
  Body fat will be measured by using Dual-emission X-ray absorptiometry
Lean body mass | Baseline
  Lean body mass will be measured by using Dual-emission X-ray absorptiometry
Dietary intake | Baseline
  Dietary intake will be assessed using 7-day diet recalls

CONTACTS AND LOCATIONS:
Overall Officials: Chariklia K Deli, PhD, Principal Investigator — Department of Physical Education and Sport Science, University of Thessaly
Locations (1):
- Department of Physical Education and Sport Science, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zafeiridis A, Saraslanidis P, Manou V, Ioakimidis P, Dipla K, Kellis S. The effects of resisted sled-pulling sprint training on acceleration and maximum speed performance. J Sports Med Phys Fitness. 2005 Sep;45(3):284-90. PMID 16230978
- [Background] Bachero-Mena B, Gonzalez-Badillo JJ. Effects of resisted sprint training on acceleration with three different loads accounting for 5, 12.5, and 20% of body mass. J Strength Cond Res. 2014 Oct;28(10):2954-60. doi: 10.1519/JSC.0000000000000492. PMID 24736770
- [Background] Baird MF, Graham SM, Baker JS, Bickerstaff GF. Creatine-kinase- and exercise-related muscle damage implications for muscle performance and recovery. J Nutr Metab. 2012;2012:960363. doi: 10.1155/2012/960363. Epub 2012 Jan 11. PMID 22288008
- [Background] Deli CK, Fatouros IG, Paschalis V, Georgakouli K, Zalavras A, Avloniti A, Koutedakis Y, Jamurtas AZ. A Comparison of Exercise-Induced Muscle Damage Following Maximal Eccentric Contractions in Men and Boys. Pediatr Exerc Sci. 2017 Aug;29(3):316-325. doi: 10.1123/pes.2016-0185. Epub 2017 Feb 6. PMID 28165870
- [Background] Petrakos G, Morin JB, Egan B. Resisted Sled Sprint Training to Improve Sprint Performance: A Systematic Review. Sports Med. 2016 Mar;46(3):381-400. doi: 10.1007/s40279-015-0422-8. PMID 26553497